CLINICAL TRIAL: NCT00070889
Title: Oxidative Cell Injury: First Episode Psychotic Patients
Brief Title: Brain Cell Injury in Patients With A First Episode of Psychosis
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: R01AT000147-01 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Psychoses
Keywords: Complementary Therapies
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Patients experiencing a first episode of psychosis may have brain cell damage due to a chemical process called oxidation. This study will compare patients with psychosis to healthy volunteers to determine if there are differences in their blood that reflect oxidative brain cell damage.

DETAILED DESCRIPTION:
Preliminary research indicated that impaired antioxidant defense and increased lipid peroxidation is associated with brain changes during the onset of psychosis. Oxidative cell injury may contribute to poor outcomes in some patients. This study will define the extent and nature of oxidative cell injury that is associated with psychopathology at the onset of psychosis.

Participants in this study will be patients at the D. D. Eisenhower Army Medical Center who are experiencing a psychotic episode for the first time. Patients will be compared with 40 healthy volunteers (control group) matched with patients for age, gender, education, ethnic background, and occupational status. Patients and volunteers will have blood tests to determine the level of oxidative cell injury. Tests will be performed at onset of psychosis, and after 6 and 12 weeks of neuroleptic drug treatment. Medical histories and MRI scans will be used to examine the relationship of the laboratory tests to the clinical presentation.

ELIGIBILITY:
Inclusion Criteria

* Patients must meet clinical diagnostic criteria for psychosis
* Healthy (control) volunteers must not have any family history of mental illness

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 1999-09; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Sahebrao P. Mahadik, PhD, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States